CLINICAL TRIAL: NCT00400426
Title: DAHANCA 20 Palliative Radiotherapy for Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Head and Neck Cancer Group (Network)
Responsible Party: Principal Investigator, Kenneth Jensen, MD ph.d., University of Aarhus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA 20
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Head and Neck Neoplasms; Recurrence; Neoplasms, Second Primary
Keywords: Palliative radiotherapy; Recurrent; Head and neck Neoplasm; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence; Neoplasms, Second Primary | interventions — Radiotherapy

INTERVENTIONS:
Procedure: Radiotherapy — 20 Gy in 4 fx

SUMMARY:
Palliative radiotherapy for head and neck cancer is widely used but the effect and side effects are largely unknown. We will study the effect of short hypofractionated palliative radiotherapy (20 Gy in 4 fractions) on symptom intensity and -frequency as weel as side effects

ELIGIBILITY:
Inclusion Criteria:

* Incurable primary or second primary head and neck cancer
* Speaks and reads Danish
* Capable of filling out questionnaires for at leas two months after radiotherapy
* Age>=18 years
* Expected survival> 3months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Frequency and intensity of symptoms before and after radiotherapy (EORTC C30 and H&N35 questionnaires and CTC AE 3.0 toxicity scores) | 11 mths

SECONDARY OUTCOMES:
Survival | 11 mths
Side effects | 2 mths
Other treatments | 11 mths

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jensen, MD, Principal Investigator — DAHANCA (Danish Head and Neck Cancer Group)
Locations (1):
- Department of Oncology, Aarhus, Denmark

REFERENCES:
- See also: Related Info — http://www.DAHANCA.dk